CLINICAL TRIAL: NCT06660745
Title: The Impact of Telenursing-based Family Empowerment Program on Self-efficacy and Treatment Adherence in Children With Cystic Fibrosis
Brief Title: The Effect of Telenursing on Self-efficacy and Treatment Adherence in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Azam Shirinabadi Farahani, Director, Correspondent Author, member of the Pediatrics Department, Principal Investigator, Associated Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IR.SBMU.PHARMACY.REC.1401.280; IRCT20230717058822N1 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis in Children
Keywords: Telenursing; Self-efficacy; Treatment adherence; Children; Cystic Fibrosis
MeSH Terms: conditions — Treatment Adherence and Compliance; Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: 50 children and adolescents with CF aged between 9-17 participated in this study.The subjects were assigned to two groups randomly, based on their medical record numbers, with even numbers placed in the intervention group and odd numbers in the control group. intervention group received twelve-week telenursing training via the SendBig website and Skype messenger and control received routine care.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group includes 25 children and their caregivers. interventional content with educational-practical and care-support model is in the form of an audio-visual file or an educational text (5-10 minutes) within a period of three months and through the content link (Send Big website) to the email address or number. It will be sent to teenager or caregiver of children with Cystic fibrosis, and after observation, remote follow-up will be done twice a week on the Skype platform, and the researcher will answer All of the questions that relate to contents. The content included topics related to various aspects of the disease and its management, Adjusting and moderating the physical activity program, medication regimen, Nutrition, and mental health.
  Interventions: Other: telenursing-based family empowerment program
- Control group (No Intervention): in control group, No intervention will take place and the patients will receive their routine treatment plan.

INTERVENTIONS:
Other: telenursing-based family empowerment program — The intervention was conducted in two sections. The first part included a one-day educational workshop conducted through Skype for the child and their caregiver and was planned to introduce the members of the intervention group to each other and provide information on how to deliver and receive the content. In the second part of the intervention, the content was prepared based on a scheduled plan. It was in the form of a 5-10-minute audio file, video, or educational text and was uploaded on the SendBig website. Once the upload is complete, a link is provided to the user. The link was sent to the phone numbers of children with cystic fibrosis and their caregivers so that they could watch the weekly content over three months. Once it was confirmed that the link had been received (acknowledged in the "Cystic Fibrosis Companions" group) and the content had been viewed, remote follow-ups were scheduled twice a week, on Sundays and Tuesdays between 6:00 PM and 8:00 PM, using Skype messenger.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if a telenursing-based programs works to increase self-efficacy and treatment adherence in children with Cystic fibrosis disease. It will also learn about the innovation and safety of this intervention.

Researchers will compare a group that received telenursing to a group with routine care to see if telenursing works to change the severity of cystic fibrosis (by changing behaviors).

Participants will be 25 in each group and were recruited during routine outpatient clinic visits in Mofid Children's Hospital during the period from April 2023 to October 2023. The participant information and consent form were provided during the first face-to-face meeting with the children and their caregivers. The patients were assigned to the intervention and control groups randomly, based on their medical record numbers, with even numbers placed in the intervention group and odd numbers in the control group. The selected communication platform (Skype) was installed by the researcher on the caregiver's and, if available, the child's mobile devices. The members of the intervention group were then added to a group called "Cystic Fibrosis Companions," which was created by the researcher on Skype. Patients in the control group continued with routine treatment and follow-up (monthly visits to the cystic fibrosis clinic and prescribed medications). For the intervention group, a telenursing-based program and follow-up were planned twice a week over twelve weeks. The intervention content for this study was derived from www.cff.org and www.cfsource.com websites and was developed by the research team. The content included topics related to various aspects of the disease and its management, Adjusting and moderating the physical activity program, medication regimen, Nutrition, and mental health. The intervention was conducted in two sections. The first part included a one-day educational workshop conducted through Skype for the child and their caregiver and was planned to introduce the members of the intervention group to each other and provide information on how to deliver and receive the content. In the second part of the intervention, the content was prepared based on a scheduled plan. It was in the form of a 5-10-minute audio file, video, or educational text and was uploaded on the SendBig website. Once the upload is complete, a link is provided to the user. The link was sent to the phone numbers of children with cystic fibrosis and their caregivers so that they could watch the weekly content over three months. Once it was confirmed that the link had been received (acknowledged in the "Cystic Fibrosis Companions" group) and the content had been viewed, remote follow-ups were scheduled twice a week, on Sundays and Tuesdays between 6:00 PM and 8:00 PM, using Skype messenger. During these sessions, the researcher reviewed the content sent that week and addressed any questions that the child and caregiver might have had about the content. These sessions also encourage interaction among the children, allow sharing of experiences gained from the interventions within each family, and allow feedback to be received. In order to prevent the control group from finding out about the content sent to the intervention group, a separate group with a different title was created on Skype, and all members of the control group were added to this new group. At the end of week 12, after the intervention was completed, the PRCISE and MATQ questionnaires were sent to the child's or caregiver's account and were completed in both control and intervention groups. Additionally, 4 weeks after the intervention, the same two questionnaires were completed again by both groups and finally, the results of the two groups were compared. At the end of the study, to observe ethical considerations, all contents were provided to the control group in the form of a compressed file containing videos, images, audio, and booklets. In this study, the mean age of the children was 12.24 in the intervention group, and 12.36 in the control group, 56% of the children with CF were boys, and 50% of them were in elementary school. A comparison of self-efficacy and treatment adherence scores indicated that the mean scores in the intervention and control groups were significantly different before and after the intervention, showing an increase immediately and one month after the intervention

ELIGIBILITY:
Inclusion Criteria:

* child's fluency in speaking, writing, and reading Farsi
* having a confirmed diagnosis of CF by a specialist
* having been diagnosed for at least one year
* not having any mental, or cognitive disorders or any other chronic diseases
* not have speech, hearing, or vision problems
* live with both parents
* have access to a smartphone
* be able to connect to the internet and send voice and text via Skype

Exclusion Criteria:

* had a Lack of interest in continuing the study
* recent pulmonary exacerbation or hospitalization during the intervention
* unable to follow educational sessions and provide feedback in at least two Q&A sessions

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Pediatric Rating of Chronic Illness Self-efficacy (PRCISE) | Before the intervention, immediately after and 4 weeks after the intervention
  The Pediatric Rating of Chronic Illness Self-Efﬁcacy scale (PRCISE) was developed by Emerson et al. (2018), to investigate the level of self-efficacy in children with chronic illnesses (20), which was reevaluated and edited by the developers in the same year and finalized with 15 items. The questionnaire was scored on an 11-point Likert scale, with zero and 150 being the minimum and maximum scores, respectively. Zero is equivalent to no self-efficacy and 150 indicates the best possible self-efficacy.

SECONDARY OUTCOMES:
The Modanloo Adherence to Treatment Questionnaire (MATQ) | Before the intervention, immediately after and 4 weeks after the intervention
  examine the level of adherence to treatment in patients with chronic disease (24), which consists of 40 items with 7 dimensions. The questionnaire was scored on a 6-point Likert scale, ranging from "Completely" with a score of 5 to "Not at all" with a score of 0. Some items are reverse-scored. The obtained scores fall between 0 and 200, and higher scores indicate better treatment adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Azam Shirinabadi Farahani, PhD, Study Director — PhD in Nursing, Associated Professor, Department of Pediatrics Nursing, School of Nursing & Midwifery, Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- Mofid Children Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The access might be possible 6 months after the results are published.
Access Criteria: The Data would be available for Researchers, students and hospital staff and it could be used for the purpose of study and research by referring to this study. the data is obtainable by Contacting with: fateme.rame@yahoo.com After sending an e-mail to the above-mentioned address in the maximum period of 1 month.